CLINICAL TRIAL: NCT02884557
Title: Evaluation of the Expression of Natural Killer T Cells (NKT) Marker in the Gut of Patients With Primary Sclerosing Cholangitis (PSC) Complicated by an Inflammatory Bowel Disease (IBD)
Brief Title: NKT Role in the Regulation of the Inflammatory Bowel Disease
Acronym: NKT-CSP/MICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011_06; 2012-A00493-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Diseases; Primary Sclerosing Cholangitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSC + IBD group (Other): collection of gut biopsies collection of blood samples in patients with PSC and IBD
  Interventions: Other: collection of gut biopsies collection of blood samples
- IBD alone group (Other): collection of gut biopsies collection of blood samples in patients with IBD alone
  Interventions: Other: collection of gut biopsies collection of blood samples

INTERVENTIONS:
Other: collection of gut biopsies collection of blood samples — Four to eight colon biopsies will be sampled during endoscopy. Thirty milliliters of blood will be sampled.

SUMMARY:
Inflammatory bowel diseases (IBD) include Crohn's disease (CD) and ulcerative colitis (UC). These diseases are a public health problem because they concern many patients (1 case in 1000). IBDs are characterized by dysregulated immune response against luminal antigens causing chronic inflammation of the gut in genetically predisposed individuals. Their exact cause is unknown and there is currently no cure. The primary sclerosing cholangitis (PSC) is a liver inflammatory disease of unknown origin that is known to be strongly associated with IBD. An important clinical observation highlights the mild symptoms of IBD when associated to the PSC. Conversely, treating PSC by liver transplant or immunosuppressive drugs is associated with a progression of intestinal inflammation.

Based, on these clinical findings that suggest a protective effect regulator of liver inflammation on intestinal inflammation, and on the results obtained by our group in mouse models that identified the natural killer T cell (NKT) as essential in control of experimental colitis, the project aims to determine, using PCR, if the expression of NKT cell markers are increased in the colon of patients with PSC+IBD compared to patients with IBD alone or PSC alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PSC alone, IBD alone or PSC + IBD
* Obtention of oral and written consent
* Patients affiliated with the social security system

Exclusion Criteria:

* Minor patient
* Suspicion of malignant lesion of the colon
* Inability for information
* person unable to consent, and not benefiting from a legal protection regimen
* Person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
The increase in the expression of the NKT marker Valpha24 mRNA by PCR in the colon of patients with PSC alone, PSC + IBD compared to patients with IBD alone | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
The number of NKT infiltrating colonic biopsies, using immunohistochemical staining | Through study completion, an average of 1 year
The percentage of NKT cells among the peripheral blood lymphocytes by flow cytometry | At the time of the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Desreumeaux, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No